CLINICAL TRIAL: NCT01073813
Title: Developing Neuroprotection and Repair Strategies in MS: Phase IIa Randomized, Controlled Trial of Minocycline in Acute Optic Neuritis (ON)
Brief Title: Neuroprotection and Repair in Optic Neuritis
Acronym: Mino in ON
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of Calgary (Other)
Collaborators: Neuroscience Canada (Unknown)
Responsible Party: Principal Investigator, Dr. Luanne Metz, Neurologist, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Minocycline in Optic Neuritis; Funding Agency (Other Grant/Funding Number: Neuroscience Canada)
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Sclerosis; Optic Neuritis
Keywords: Minocycline; Retinal nerve fibre layer thickness; Macular volume; Visual outcomes
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minocycline 100mg (Active Comparator): Patients are in one of three strata (currently on Glatiramer acetate (GA), Interferon beta (IFN), or neither disease modifying therapy (DMT). There will be a minimum of 12 patients per strata. Patients will be randomized within each strata in a 2:1 fashion to receive either Minocycline 100mg twice daily or no treatment.
  Interventions: Drug: Minocycline
- No treatment (No Intervention): Patients are in one of three strata (currently on Glatiramer acetate (GA), Interferon beta (IFN), or neither disease modifying therapy (DMT). There will be a minimum of 12 patients per strata. Patients will be randomized within each strata in a 2:1 fashion to receive either Minocycline 100mg twice daily or no treatment.

INTERVENTIONS:
Drug: Minocycline — 100mg twice daily
  Arms: Minocycline 100mg

SUMMARY:
The primary aim of this open-label pilot trial is to estimate the treatment effect of 100 mg of oral minocycline twice daily for 90 days, initiated within 30 days of onset of ON, on functional and structural optic nerve recovery compared to no treatment. The primary outcome measure that will be used to measure optic nerve recovery is retinal nerve fibre layer (RNFL) thickness. Other objectives: Secondary outcomes are temporal RNFL thickness, macular volume, and visual outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years, the lower age limit has been set for safety purposes to avoid exposing children and adolescents to unproven therapies at least early in their development, the upper limit is set because the specificity of the diagnosis of ON is likely reduced in older individuals
* onset of ON within the previous 30 days
* intention to continue current multiple sclerosis (MS) disease modifying therapy (if any) for at least 6 months (glatiramer acetate, interferon beta) and not start, or switch to, a new therapy
* sexually active participants of child-bearing potential must agree to use adequate contraception
* willingness to provide written informed consent

Exclusion Criteria:

* Coexistence of any disease other than MS that could be responsible for ON or better explains their signs and symptoms. This would include patients with other suspected or established causes of vision loss including glaucoma, maculopathies, amblyopia, neuro-myelitis optica (NMO), and other optic neuropathies
* clinically significant liver, renal, or bone marrow dysfunction
* any condition that could interfere with any evaluation in the study including patients who are unable to undergo reliable OCT testing due to dense media opacities or severe nystagmus in whom appropriate fixation cannot be attained
* concurrent or prior use of corticosteroids during this episode of optic neuritis
* concurrent participation in any clinical therapeutic trial
* use within the previous 12 months of any of the following: natalizumab, mitoxantrone, cyclophosphamide, azathioprine, cyclosporine, methotrexate, or any other immunomodulating or immunosuppressive drug including other recombinant or non-recombinant cytokine or any experimental therapy known to effect immune function
* use within the previous 6 months of minocycline or another tetracycline or use of either for MS at any time
* any other condition or situation that in the opinion of the investigator would either put the patient at risk of worsening health if enrolled in the trial or would prevent completion of the trial with complete follow-up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Retinal nerve fibre layer | At baseline and every three months for nine months
  The primary aim of this open-label pilot trial is to estimate the treatment effect of 100 mg of oral minocycline twice daily for 90 days, initiated within 30 days of onset of ON, on functional and structural optic nerve recovery compared to no treatment. The primary outcome measure that will be used to measure optic nerve recovery is RNFL thickness.

SECONDARY OUTCOMES:
Other functional and structural optic nerve recovery measures | At baseline and every three months for nine months
  Secondary outcomes are temporal RNFL thickness, macular volume, and visual outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Luanne Metz, Dr., Principal Investigator — University of Calgary; Fiona Costello, Dr., Principal Investigator — University of Calgary